CLINICAL TRIAL: NCT01075711
Title: Non-interventional Study for Determining the Improvement in the Activity Status / Life Quality of Patients With Rheumatoid Arthritis Being Treated With the Tempus Tablet
Brief Title: Determine the Improvement in Activity Status/Quality of Life (QoL) of Patients With Rheumatoid Arthritis (RA) During Treatment With Lodotra (Prednisone)
Acronym: LODOTRA
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono GmbH, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 062215-500
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Prednisone
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample

GROUPS / COHORTS (2):
- NIS in-house doctors: This group will be assigned to general physicians, practicing doctors and interns (in-house doctors) with an observation period of 3 months. Three subjects are expected per in-house doctor therefore altogether, 1000 in-house doctors will be obtained or appointed for the observation study.
  Interventions: Drug: Prednisone
- NIS specialists: This group will be assigned to specialists (rheumatologist) with an observation period of 9 months. Ten subjects per rheumatologist are expected therefore altogether, 500 rheumatologists will be obtained or appointed for the observation study.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — According to SPC
  Other Names: Lodotra

SUMMARY:
Rheumatoid arthritis is the most common rheumatic disease with symptomatic morning stiffness which entails a quite essential restriction in the everyday life and in the life quality. This observational, uncontrolled, multicentric study is aimed to assess the improvement in the activity status or QoL of subjects with RA being treated with the Tempus tablet.

DETAILED DESCRIPTION:
Rheumatoid arthritis is characterised with a sudden onset , with pains in the little finger or toe joints, progressively affecting various joints and symptomatic morning stiffness. For subjects with RA, morning stiffness entails a quite essential restriction in the everyday life and in the life quality. This observational, uncontrolled, multicentric study is aimed to assess the improvement in the activity status or QoL of subjects with RA being treated with the Tempus tablet. A total of 8,000 subjects with diagnosed, active RA will be included in the study The study will apply to 2 target groups: general physicians, practicing doctors and interns (in-house doctors) with an observation period of 3 months; and specialists (rheumatologist) with an observation period of 9 months. Three subjects are expected per in-house doctor and 10 subjects per rheumatologist.

OBJECTIVES

Primary Objective:

* To examine, to what extent the subject will be directly benefited with the decrease in the morning arthritis symptom in the sense of an improvement in the life quality and the activity status

  1. The activity status will be assessed in 3 different areas: occupational activities, tasks in the household and leisure activities
  2. The life quality is assessed on the basis of the HAQ-DI

Secondary Objectives:

* To record side effects of Tempus tablet when used under everyday conditions
* To collect socioeconomic data such as e.g. aids or applications

ELIGIBILITY:
Inclusion Criteria:

* Subjects who correspond to the permitted indication of the drug of Lodotra
* Subjects from age of 18 years with diagnosed, active RA with associated symptoms such as morning stiffness of the joints, which is either already being treated with low dose of glucocorticoids or will be treated again with glucocorticoid therapy

Exclusion Criteria:

* - Subjects with contraindications are excluded from the participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with RA who are treated with Tempus tablet and subjects with re-diagnosed RA are also included in the study, if the RA is treated with glucocorticoides.
Sampling Method: Probability Sample
Enrollment: 2728 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in the QAS (Questionnaire on Activity Status) | Beginning of the examination (gross-root survey) and after 3 months (follow-up)

SECONDARY OUTCOMES:
QAS comparison after 9 months | Beginning until after 9 months
Performance by visual analog scale (VAS) | Beginning until after 9 months
Concurrent medication | Beginning until after 9 months
Health Assessment Questionnaire Disability Index (HAQ-DI) (NIS specialists) | Beginning until after 9 months
Laboratory results (c reactive protein [CRP], BSG), X-rays (if available) | Beginning until after 9 months
Side-effects and undesirable events | Beginning until after 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Boris Pfeiffer, M.Sc., Study Director — Merck Serono GmbH, Germany
Locations (1):
- Merck Serono GmbH, Darmstadt, Germany, Darmstadt, Germany

REFERENCES:
- [Result] Pfeiffer BM, Krenzer S, Dockhorn R, Schwenke R, Schwenke H, Waehrisch J, Kraus E. Impact of modified-release prednisone on functional ability in patients with rheumatoid arthritis. Rheumatol Int. 2013 Jun;33(6):1447-54. doi: 10.1007/s00296-012-2583-1. Epub 2012 Nov 21. PMID 23179262